CLINICAL TRIAL: NCT02721732
Title: Phase II Study for the Evaluation of Efficacy of Pembrolizumab (MK-3475) in Patients With Rare Tumors
Brief Title: Pembrolizumab in Treating Patients With Rare Tumors That Cannot Be Removed by Surgery or Are Metastatic
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0948; NCI-2016-00545 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0948 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Results first posted 2024-06-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Carcinoma of Unknown Primary; Metastatic Adrenal Gland Pheochromocytoma; Metastatic Kidney Medullary Carcinoma; Metastatic Malignant Germ Cell Tumor; Metastatic Malignant Solid Neoplasm; Metastatic Paraganglioma; Metastatic Penile Carcinoma; Metastatic Skin Squamous Cell Carcinoma; Small Cell Carcinoma; Stage III Adrenal Cortex Carcinoma AJCC v7; Stage IV Adrenal Cortex Carcinoma AJCC v7; Stage IV Penile Cancer AJCC v7; Stage IV Renal Cell Cancer AJCC v7; Unresectable Adrenal Gland Pheochromocytoma; Unresectable Paraganglioma; Unresectable Skin Squamous Cell Carcinoma; Unresectable Solid Neoplasm; Vascular Neoplasm
MeSH Terms: conditions — Neoplasms, Unknown Primary; Pheochromocytoma; Neoplasm Metastasis; Paraganglioma; Penile Neoplasms; Carcinoma, Small Cell; Adrenal Cortex Neoplasms; Carcinoma, Renal Cell; Vascular Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression or toxicity. Patients with clinical response or disease stabilization may continue treatment for up to an additional 12 months.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with rare tumors that cannot be removed by surgery or have spread to other parts of the body. Monoclonal antibodies, such as pembrolizumab, may block specific proteins found on white blood cells which may strengthen the immune system and control tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain early indication of efficacy by evaluation of non-progression rate (NPR) at 27 weeks as defined as the percentage of patients who are alive and progression-free at 27 weeks as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 or immune-related(ir)RECIST or method of tumor evaluation criteria best suitable and accepted for the tumor type evaluated in patients with advanced tumor types receiving pembrolizumab.

SECONDARY OBJECTIVES:

I. To correlate efficacy by evaluation of tumor size to programmed cell death 1 ligand 1 (PD-L1) status among patients with advanced tumor types receiving pembrolizumab.

II. To evaluate safety and tolerability of pembrolizumab in patients with advanced tumors.

III. To evaluate the percentage of patients with objective response (complete response [CR] or partial response [PR]), clinical benefit (CR, PR, or stable disease [SD] >= 4 months), progression free survival (PFS), overall survival (OS), and duration of response (DOR) as assessed by RECIST v1.1 in patients with advanced tumor types receiving pembrolizumab.

IV. To evaluate the percentage of patients with objective response (CR or PR), clinical benefit (CR, PR, or SD >= 4 months), PFS, and DOR as assessed by irRECIST in patients with advanced tumor types receiving pembrolizumab.

V. To correlate the NPR at 27 weeks (9 cycles), objective response (CR or PR), clinical benefit CR, PR, or SD >= 4 months), PFS, OS, and DOR to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.

EXPLORATORY OBJECTIVES:

I. To evaluate the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness in patients with advanced tumor types receiving pembrolizumab.

II. To correlate the potential role of tumor-associated immune biomarkers for prediction of therapy effectiveness to PD-L1 status among patients with advanced tumor types receiving pembrolizumab.

III. To identify imaging characteristics associated with immunological changes in tumor following treatment with pembrolizumab.

IV. To compare tumor mutation burden and serial assessment of mutation status in biopsies obtained at baseline and progression in patients with advanced tumor types receiving pembrolizumab.

V. To evaluate patient-reported outcomes (PRO) utilizing the National Cancer Institute (NCI) Patient-Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) questionnaires.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 24 months in the absence of disease progression or toxicity. Patients with clinical response or disease stabilization may continue treatment for up to an additional 12 months.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease based on RECIST 1.1 or irRECIST; only cohort 9 and 10 can have evaluable disease (non-measurable lesions); tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions; patients may have bone metastatic disease evaluable according to tumor evaluation criteria best suitable and accepted for the tumor type evaluated
* Have one of the following advanced (unresectable and/or metastatic) solid tumor indications that has progressed following standard therapies, where standard therapies are available:

  * Squamous cell carcinoma of the skin
  * Small cell malignancies of non-pulmonary origin
  * Adrenocortical carcinoma
  * Medullary renal cell carcinoma
  * Carcinoma of unknown primary
  * Penile carcinoma
  * Vascular sarcoma
  * Germ cell tumor
  * Paraganglioma-pheochromocytoma
  * Other rare tumors (except those tumor types listed in exclusion)
* Have failed prior treatment within 6 months of consent date
* Have biopsiable disease; subjects must have at least one lesion amenable to biopsy; tumor lesions used for biopsy should not be lesions used as target lesions; in cohort 9: paraganglioma-pheochromocytoma or cohort 10, where there is prominent bony disease, biopsies may not be possible due to the nature of the disease
* Be willing to provide archival tissue; if archival tissue is not available, or a newly obtained core or excisional biopsy of a tumor lesion will be obtained; newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1; in cohort 9: paraganglioma-pheochromocytoma or cohort 10, where there is prominent bony disease, biopsies may not be possible due to the nature of the disease
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,000/mcL (performed within 28 days of treatment initiation)
* Platelets >= 75,000/mcL (performed within 28 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (performed within 28 days of treatment initiation)
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (performed within 28 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 28 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (performed within 28 days of treatment initiation)
* Albumin > 2.5 mg/dL (performed within 28 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 28 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 28 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* For subjects in cohort 2 (small cell malignancies of non-pulmonary origin), confirmation of no brain metastases via imaging

Exclusion Criteria:

* Is currently participating and receiving study therapy or concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment at the time of administration of first dose of trial treatment; continuation of hormone replacement therapy is permitted; stable regimens of hormonal therapy i.e. for prostate cancer (e.g. leuprolide, a gonadotrophin releasing hormone [GnRH] agonist), ovarian, or breast cancer are not exclusionary
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent; Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study; Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer, and diseases for which the treatment could reasonably include pembrolizumab and are not part of the excluded tumor type list or not eligible for the phase I trial
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; immunosuppressive corticosteroid doses (> 10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of pembrolizumab; Note: corticosteroids given within 24 hours of an imaging study for purposes of pre-medication in patients with hypersensitivity to radiologic contrast agents are allowed
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Is participating in cohort 10 and has melanoma; non-small cell lung cancer; hepatocellular carcinoma; Merkel cell carcinoma; colon or rectal adenocarcinoma; anal canal squamous cell carcinoma; pancreas adenocarcinoma; esophageal squamous cell carcinoma or adenocarcinoma (including gastroesophageal [GE] junction); biliary tract adenocarcinoma (gallbladder and biliary tree but excluding ampulla of vater cancers); carcinoid tumors; neuroendocrine carcinomas (well or moderately differentiated pancreatic neuroendocrine tumor); estrogen receptor (ER)-positive human epidermal growth factor receptor 2 (HER2)-negative breast cancer; triple negative breast cancer; ovarian epithelial, fallopian tube or primary peritoneal carcinoma; endometrial carcinoma; cervical squamous cell cancer; vulvar squamous cell carcinoma; small cell lung cancer; mesothelioma (malignant pleural mesothelioma); thyroid cancer (papillary or follicular subtype); salivary gland carcinoma; nasopharyngeal carcinoma; glioblastoma multiforme; leiomyosarcoma; prostate adenocarcinoma; gastric adenocarcinoma; or small bowel malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chahla B, Stephen B, Song J, Balderrama-Brondani V, Yaylaci F, Campbell MT, Naing A, Habra MA. Phase 2 Study of Monotherapy with Pembrolizumab for Advanced Adrenocortical Carcinoma. J Immunother Precis Oncol. 2025 Oct 6;8(4):242-248. doi: 10.36401/JIPO-25-6. eCollection 2025 Nov. PMID 41143139
- [Derived] Nardo M, Braganca Xavier C, Stephen B, How JA, Moyers J, Subbiah V, Hong DS, Naing A. Pembrolizumab in Patients with Advanced Miscellaneous Rare Cancers: Results from a Phase 2 Basket Trial. J Immunother Precis Oncol. 2025 Apr 10;8(2):143-151. doi: 10.36401/JIPO-24-27. eCollection 2025 May. PMID 40212844
- [Derived] Nze C, Msaouel P, Derbala MH, Stephen B, Abonofal A, Meric-Bernstam F, Tannir NM, Naing A. A Phase II Clinical Trial of Pembrolizumab Efficacy and Safety in Advanced Renal Medullary Carcinoma. Cancers (Basel). 2023 Jul 27;15(15):3806. doi: 10.3390/cancers15153806. PMID 37568622
- [Derived] Mendoza TR, Hong DS, Peterson CB, Stephen B, Dumbrava E, Pant S, Tsimberidou AM, Yap TA, Sheshadri A, Altan M, George G, Castillo L, Rodriguez E, Gong J, Subbiah V, Janku F, Fu S, Piha-Paul SA, Ahnert JR, Karp DD, Cleeland C, Meric-Bernstam F, Naing A. Patient-reported symptom burden in patients with rare cancers receiving pembrolizumab in a phase II Clinical Trial. Sci Rep. 2022 Aug 23;12(1):14367. doi: 10.1038/s41598-022-16588-3. PMID 35999229
- [Derived] Raghav KP, Stephen B, Karp DD, Piha-Paul SA, Hong DS, Jain D, Chudy Onwugaje DO, Abonofal A, Willett AF, Overman M, Smaglo B, Huey RW, Meric-Bernstam F, Varadhachary GR, Naing A. Efficacy of pembrolizumab in patients with advanced cancer of unknown primary (CUP): a phase 2 non-randomized clinical trial. J Immunother Cancer. 2022 May;10(5):e004822. doi: 10.1136/jitc-2022-004822. PMID 35618285
- [Derived] Pant S, Moyers JT, Naing A. Letter to the editor from Pant et al. J Immunother Cancer. 2021 Nov;9(11):e003991. doi: 10.1136/jitc-2021-003991. No abstract available. PMID 34725215
- [Derived] Ferrarotto R, Sousa LG, Qing Y, Kaya D, Stephen B, Jain D, Bell D, Pant S, Tsimberidou AM, Janku F, Blumenschein G, Glisson BS, Ahnert JR, Piha-Paul SA, Lee JJ, Wong MK, Lu C, Meric-Bernstam F, Naing A. Pembrolizumab in Patients with Refractory Cutaneous Squamous Cell Carcinoma: A Phase II Trial. Adv Ther. 2021 Aug;38(8):4581-4591. doi: 10.1007/s12325-021-01807-6. Epub 2021 Jul 9. PMID 34241781
- [Derived] Hahn AW, Chahoud J, Campbell MT, Karp DD, Wang J, Stephen B, Tu SM, Pettaway CA, Naing A. Pembrolizumab for advanced penile cancer: a case series from a phase II basket trial. Invest New Drugs. 2021 Oct;39(5):1405-1410. doi: 10.1007/s10637-021-01100-x. Epub 2021 Mar 26. PMID 33770291
- [Derived] Tsimberidou AM, Vo HH, Subbiah V, Janku F, Piha-Paul S, Yilmaz B, Gong J, Naqvi MF, Tu SM, Campbell M, Meric-Bernstam F, Naing A. Pembrolizumab in Patients with Advanced Metastatic Germ Cell Tumors. Oncologist. 2021 Jul;26(7):558-e1098. doi: 10.1002/onco.13682. Epub 2021 Feb 12. PMID 33491277
- [Derived] Majd N, Waguespack SG, Janku F, Fu S, Penas-Prado M, Xu M, Alshawa A, Kamiya-Matsuoka C, Raza SM, McCutcheon IE, Naing A. Efficacy of pembrolizumab in patients with pituitary carcinoma: report of four cases from a phase II study. J Immunother Cancer. 2020 Dec;8(2):e001532. doi: 10.1136/jitc-2020-001532. PMID 33427689
- [Derived] How JA, Jazaeri A, Westin SN, Sood AK, Ramondetta LM, Xu M, Abonofal A, Karp DD, Subbiah V, Stephen B, Rodon JA, Yang F, Naing A. The clinical efficacy and safety of single-agent pembrolizumab in patients with recurrent granulosa cell tumors of the ovary: a case series from a phase II basket trial. Invest New Drugs. 2021 Jun;39(3):829-835. doi: 10.1007/s10637-020-01043-9. Epub 2021 Jan 7. PMID 33415580
- [Derived] Frumovitz M, Westin SN, Salvo G, Zarifa A, Xu M, Yap TA, Rodon AJ, Karp DD, Abonofal A, Jazaeri AA, Naing A. Phase II study of pembrolizumab efficacy and safety in women with recurrent small cell neuroendocrine carcinoma of the lower genital tract. Gynecol Oncol. 2020 Sep;158(3):570-575. doi: 10.1016/j.ygyno.2020.05.682. Epub 2020 Jun 11. PMID 32534809
- [Derived] Tapia C, Aung PP, Roy-Chowdhuri S, Xu M, Ouyang F, Alshawa A, Hajjar J, Singh G, Yang V, Castillo L, Le H, Murthy R, Stephen B, Hess KR, Wistuba I, Naing A. Decrease in tumor content assessed in biopsies is associated with improved treatment outcome response to pembrolizumab in patients with rare tumors. J Immunother Cancer. 2020 Apr;8(1):e000665. doi: 10.1136/jitc-2020-000665. PMID 32303619
- [Derived] Naing A, Meric-Bernstam F, Stephen B, Karp DD, Hajjar J, Rodon Ahnert J, Piha-Paul SA, Colen RR, Jimenez C, Raghav KP, Ferrarotto R, Tu SM, Campbell M, Wang L, Sabir SH, Tapia C, Bernatchez C, Frumovitz M, Tannir N, Ravi V, Khan S, Painter JM, Abonofal A, Gong J, Alshawa A, McQuinn LM, Xu M, Ahmed S, Subbiah V, Hong DS, Pant S, Yap TA, Tsimberidou AM, Dumbrava EEI, Janku F, Fu S, Simon RM, Hess KR, Varadhachary GR, Habra MA. Phase 2 study of pembrolizumab in patients with advanced rare cancers. J Immunother Cancer. 2020 Mar;8(1):e000347. doi: 10.1136/jitc-2019-000347. PMID 32188704
- [Derived] Habra MA, Stephen B, Campbell M, Hess K, Tapia C, Xu M, Rodon Ahnert J, Jimenez C, Lee JE, Perrier ND, Boraddus RR, Pant S, Subbiah V, Hong DS, Zarifa A, Fu S, Karp DD, Meric-Bernstam F, Naing A. Phase II clinical trial of pembrolizumab efficacy and safety in advanced adrenocortical carcinoma. J Immunother Cancer. 2019 Sep 18;7(1):253. doi: 10.1186/s40425-019-0722-x. PMID 31533818
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single-center, open-label, phase II trial of pembrolizumab (MK-3475) in patients with and without programmed death-ligand 1 (PD-L1) positive advanced tumors conducted at the University of Texas MD Anderson Cancer Center
Groups:
- Cohort 1: Squamous Cell Carcinoma of the Skin; Cohort 2: Small Cell Malignancies of Nonpulmonary Origin; Cohort 3: Adrenocortical Carcinoma; Cohort 4: Medullary Renal Cell Carcinoma; Cohort 5: Carcinoma of Unknown Primary; Cohort 6: Penile Carcinoma; Cohort 7: Vascular Sarcoma; Cohort 8: Germ Cell Tumor; Cohort 9: Paraganglioma-pheochromocytoma; Cohort 10: Other Rare Tumor Histologies: MK-3475: 200 mg of MK-3475 administered intravenously on Day 1 of every 21-day cycle
Period: Overall Study
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Started | 20 | 12 | 24 | 5 | 29 | 3 | 11 | 12 | 13 | 28
Completed | 3 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 2 | 3
Not Completed | 17 | 12 | 22 | 5 | 26 | 3 | 11 | 12 | 11 | 25
Not completed — Adverse Event | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 12 | 11 | 18 | 5 | 21 | 2 | 8 | 11 | 10 | 20
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 1
Not completed — Participant Choice | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progression and Exclusion from study due to changed diagnosis | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progression and withdrew consent | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — No evidence of tumor following radical surgery | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies | Total
Number analyzed (Participants) | 20 | 12 | 24 | 5 | 29 | 3 | 11 | 12 | 13 | 28 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 10 | 20 | 5 | 15 | 0 | 5 | 12 | 12 | 21 | 106
  >=65 years | 14 | 2 | 4 | 0 | 14 | 3 | 6 | 0 | 1 | 7 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 14 | 1 | 21 | 0 | 4 | 2 | 5 | 19 | 76
  Male | 17 | 5 | 10 | 4 | 8 | 3 | 7 | 10 | 8 | 9 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 0 | 2 | 1 | 0 | 3 | 2 | 4 | 16
  Not Hispanic or Latino | 20 | 9 | 22 | 5 | 25 | 2 | 11 | 9 | 11 | 24 | 138
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 3 | 3 | 0 | 0 | 1 | 1 | 3 | 12
  White | 20 | 10 | 19 | 1 | 22 | 2 | 8 | 8 | 10 | 18 | 118
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 3 | 0 | 2 | 3 | 2 | 5 | 18
Region of Enrollment [Number; unit: participants]
  United States | 20 | 12 | 24 | 5 | 29 | 3 | 11 | 12 | 13 | 28 | 157

OUTCOME MEASURES:

1. Primary Outcome: Non-progression Rate (NPR) at 27 Weeks by irRECIST
Description: Non-progression rate (NPR) at 27 weeks was defined as the percentage of efficacy evaluable patients who were alive and progression-free at 27 weeks as assessed by irRECIST
  Progression is defined using immune-related Response Evaluation Criteria in Solid Tumors (irRECIST), as an increase ≥ 20% (minimum 5 mm) in total measured tumor burden compared with nadir or progression of non-target lesions or new lesion
Time Frame: At 27 weeks
Population: All patients who have received at least 1 dose of study medication with at least 1on-study tumor assessment were included in the analysis. If a patient discontinued before the first radiological assessment due to progression, they were included in the analysis. If the patient discontinued before 27 weeks due to reasons other than progression or death, they were considered non evaluable for this endpoint. One patient enrolled in the ACC cohort was excluded due to change in diagnosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Number analyzed (Participants) | 17 | 12 | 20 | 5 | 26 | 2 | 10 | 11 | 12 | 27
Participants | 7 | 0 | 6 | 0 | 8 | 0 | 2 | 1 | 4 | 9

2. Secondary Outcome: Evaluation of Tumor Size (Objective Response by irRECIST) to PD-L1 Status (CPS ≥1)
Description: Immune-related ORR is defined as the percentage of patients achieving a irCR or irPR based on irRECIST criteria. PD-L1 positivity was defined as Combined Positive Score ≥1. Evaluated objective response in PD-L1 positive patients
  Per irRECIST: Immune-related (ir) Complete Response (irCR), disappearance of all target and non-target lesions, nodal short axis diameter <10 mm, no new lesions; irPartial Response (irPR), decrease of ≥30% in tumor burden relative to baseline, non-unequivocal progression of non-target lesions, no new lesions.
Time Frame: Baseline and every 9 weeks thereafter. After 6 months, every 12 weeks at the physician's discretion, if patient has had CR, PR, or SD > 27 weeks, an average of 4 years.
Population: PD-L1 expression on tumor and mononuclear inflammatory cells in tumor nests were assessed on samples obtained prior to treatment. Patients with PD-L1 positive disease (CPS ≥1) were evaluated for objective response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Number analyzed (Participants) | 14 | 6 | 2 | 4 | 16 | 2 | 6 | 3 | 5 | 14
Participants | 6 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 1

3. Secondary Outcome: Number of Patients Who Experienced Treatment-related Adverse Event (TRAE)
Description: Per protocol, the number and percentage of patients with any treatment-related AE was summarized for all study patients combined. Patients were monitored for AE from the first day of administration of study medication through 30 days following last dose. Each AE (as defined by NCI CTCAE v4.03) was counted only once for a given subject. In the event a patient experienced repeated episodes of the same AE, then the event with the highest severity and/or strongest causal relationship to study treatment was used for purposes of tabulations.
Time Frame: First day of administration of study medication through 30 days following last dose, an average of 4 years.
Population: It was a pre-specified objective. All patients who have received at least 1 dose of study medication were included in the safety analysis. A total of 157 patients were treated on this study. One patient enrolled in the ACC cohort was excluded from the study due to change in the diagnosis following histological assessment of the surgical specimen.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients Who Received at Least One Dose of the Drug: MK-3475: 200 mg of MK-3475 administered intravenously on Day 1 of every 21-day cycle
Arm/Group | All Patients Who Received at Least One Dose of the Drug
Number analyzed (Participants) | 156
Participants | 88

4. Secondary Outcome: Objective Response Rate (ORR) Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: ORR is defined as the percentage of patients achieving a complete response (CR) or partial response (PR) based on RECIST 1.1 criteria.
Time Frame: as for outcome 2
Population: All patients who have received at least 1 dose of study medication with at least one adequate on-study tumor assessment were included in the efficacy analysis. If a patient discontinued the study before the first radiological assessment due to progression of disease, either radiological or clinical, they were considered evaluable and were included in the efficacy analysis. One patient enrolled in the ACC cohort was excluded from the study due to change in the diagnosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Number analyzed (Participants) | 18 | 12 | 20 | 5 | 26 | 3 | 10 | 11 | 13 | 28
Participants | 6 | 0 | 4 | 0 | 5 | 1 | 1 | 0 | 1 | 5

5. Secondary Outcome: Clinical Benefit Rate (CBR) Using RECIST v1.1
Description: CBR is defined as the percentage of patients achieving a CR or PR, or stable disease (SD) ≥4 months based on RECIST 1.1 criteria.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Number analyzed (Participants) | 18 | 12 | 20 | 5 | 26 | 3 | 10 | 11 | 13 | 28
Participants | 7 | 0 | 11 | 0 | 10 | 1 | 3 | 2 | 7 | 13

6. Secondary Outcome: Progression-free Survival (PFS) Using RECIST v1.1
Description: PFS was defined as the time from administration of the first dose to the first documented disease progression according to RECIST v1.1 or death due to any cause, whichever occurs first. Patients who were alive and had not experienced disease progression at the time of data cutoff were censored.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients Who Received at Least One Dose of the Drug
Number analyzed (Participants) | 146
months | 2.2 [2 to 2.7]

7. Secondary Outcome: Immune-related ORR Using Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: Immune-related ORR is defined as the percentage of patients achieving a irCR or irPR based on irRECIST criteria.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Number analyzed (Participants) | 18 | 12 | 20 | 5 | 26 | 3 | 10 | 11 | 13 | 28
Participants | 6 | 0 | 4 | 0 | 5 | 1 | 1 | 0 | 1 | 5

8. Secondary Outcome: Immune-related Clinical Benefit Rate (CBR) Using irRECIST
Description: Immune-related CBR is defined as the percentage of patients achieving a irCR or irPR, or irSD ≥4 months based on irRECIST criteria
Time Frame: First day of administration of study medication through 30 days following last dose, an average of 4 years.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Squamous Cell Carcinoma of the Skin | Cohort 2: Small Cell Malignancies of Nonpulmonary Origin | Cohort 3: Adrenocortical Carcinoma | Cohort 4: Medullary Renal Cell Carcinoma | Cohort 5: Carcinoma of Unknown Primary | Cohort 6: Penile Carcinoma | Cohort 7: Vascular Sarcoma | Cohort 8: Germ Cell Tumor | Cohort 9: Paraganglioma-pheochromocytoma | Cohort 10: Other Rare Tumor Histologies
Number analyzed (Participants) | 18 | 12 | 20 | 5 | 26 | 3 | 10 | 11 | 13 | 28
Participants | 8 | 0 | 11 | 0 | 12 | 1 | 3 | 2 | 7 | 14

9. Secondary Outcome: Immune-related Progression-free Survival (PFS) Using irRECIST
Description: Immune-related PFS was defined as the time from administration of the first dose to the first documented disease progression according to irRECIST or death due to any cause, whichever occurs first. Patients who were alive and had not experienced disease progression at the time of data cutoff were censored.
Time Frame: Baseline and every 9 weeks thereafter. After 6 months, every 12 weeks at the physician's discretion, if patient has had CR, PR, or SD > 27 weeks.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients Who Received at Least One Dose of the Drug
Number analyzed (Participants) | 146
months | 2.3 [2 to 3.6]

ADVERSE EVENTS:
Time Frame: First day of administration of study medication through 30 days following last dose.
Description: All participants received the same intervention. Therefore, per protocol, all cause-mortality, SAEs and other AEs are reported for all study patients combined.
Groups:
- Participants With Advanced Rare Cancer: "MK-3475: 200 mg IV on Day 1 of every 21-day cycle Of the 157 participants enrolled, one participant in ACC cohort was excluded due to change in the diagnosis."
Arm/Group | Participants With Advanced Rare Cancer
All-Cause Mortality (participants affected / at risk) | 114/156
Serious Adverse Events (participants affected / at risk) | 72/156
Other Adverse Events (participants affected / at risk) | 84/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Advanced Rare Cancer (N=156)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Fever (General disorders) | 5 (5)
Lung infection (Infections and infestations) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Hematoma (Vascular disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Autoimmune disorder (hepatitis) (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
NOS, Neoplasms benign,malignant and unspecified (incl cysts and polyps) -Other, (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasms benign,malignant and unspecified (incl cysts and polyps) -Other, specify-Tumor bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify-Altered mental (Psychiatric disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal and urinary disorders - Other, specify-acute renal failure (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Advanced Rare Cancer (N=156)
Fatigue (General disorders) | 55 (55)
Anemia (Blood and lymphatic system disorders) | 52 (52)
Constipation (Gastrointestinal disorders) | 41 (41)
Creatinine increased (Investigations) | 35 (35)
Aspartate aminotransferase increased (Investigations) | 32 (32)
Alanine aminotransferase increased (Investigations) | 31 (31)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 (31)
Alkaline phosphatase increased (Investigations) | 28 (28)
Nausea (Gastrointestinal disorders) | 28 (28)
Hypothyroidism (Endocrine disorders) | 27 (27)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 (26)
Hyperglycemia (Metabolism and nutrition disorders) | 25 (25)
Anorexia (Metabolism and nutrition disorders) | 24 (24)
Diarrhea (Gastrointestinal disorders) | 24 (24)
Hypomagnesemia (Metabolism and nutrition disorders) | 24 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 22 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (21)
Hyperuricemia (Metabolism and nutrition disorders) | 18 (18)
Hyponatremia (Metabolism and nutrition disorders) | 16 (16)
Hypercalcemia (Metabolism and nutrition disorders) | 14 (14)
Headache (Nervous system disorders) | 13 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (13)
Platelet count decreased (Investigations) | 13 (13)
Edema limbs (General disorders) | 12 (12)
Pain (General disorders) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 10 (10)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 10 (10)
Upper respiratory infection (Infections and infestations) | 10 (10)
Abdominal pain (Gastrointestinal disorders) | 9 (9)
Fever (General disorders) | 9 (9)
Hypotension (Vascular disorders) | 9 (9)
Insomnia (Psychiatric disorders) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 9 (9)
White blood cell decreased (Investigations) | 9 (9)
Activated partial thromboplastin time prolonged (Investigations) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
General disorders and administration site conditions - Other, specify (General disorders) | 8 (8)
Blood bilirubin increased (Investigations) | 7 (7)
Hypertension (Vascular disorders) | 7 (7)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Hyperthyroidism (Endocrine disorders) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
Investigations - Other, specify (Investigations) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Lymphocyte count decreased (Investigations) | 5 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 5 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Endocrine disorders - Other, specify (Endocrine disorders) | 4 (4)
Eye disorders - Other, specify (Eye disorders) | 4 (4)
INR increased (Investigations) | 4 (4)
Lung infection (Infections and infestations) | 4 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (4)
Neutrophil count decreased (Investigations) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Blurred vision (Eye disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Localized edema (General disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Vaginal infection (Infections and infestations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Hair loss to armpits and legs (General disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased PTT (Investigations) | 1 (1)
Increased Prothrombin time (Investigations) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg swelling (General disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Poor appetite (Metabolism and nutrition disorders) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Testicular disorder (Reproductive system and breast disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT02721732/Prot_SAP_000.pdf